CLINICAL TRIAL: NCT07398781
Title: The PACE Study (Present-Moment Awareness, Attention, Compassion, Emotion Regulation): Effects of a School-Based Mindfulness and Compassion Intervention
Brief Title: PACE Study: A School-Based Mindfulness and Compassion Intervention in Children
Acronym: PACE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Pisa (Other); University of Florence (Other); John Cabot University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PACE
Record Dates: First submitted 2026-01-05; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: School-based Intervention; Mindfulness-based Intervention; Compassion; Emotion Regulation
Keywords: mindfulness; compassion; emotion regulation; School
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PACE intervention (Experimental): Children in this arm will participate in the PACE program, a school-based intervention consisting of structured activities focused on mindfulness, compassion, and emotion regulation.
  Interventions: Behavioral: Mindfulness-based intervention

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The PACE intervention is a five-session, school-based program aimed at improving students' mindfulness, self-compassion, and emotion regulation. Assessments of attention, executive functions, mindfulness, and emotional well-being are conducted before and after the intervention.

SUMMARY:
This study aims to evaluate the effects of a school-based intervention grounded in mindfulness, compassion, and emotion regulation on children's psychological well-being and higher-order cognitive functions.

The intervention is delivered in a classroom setting through structured experiential activities. Children are assessed before and after the intervention using standardized tests and questionnaires measuring attention, executive functions, emotional regulation, mindfulness, and self-compassion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be primary school students (age 6-11)

Exclusion Criteria:

* Lack of signed consent

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mindfulness | 10 days before intervention and 10 days after intervention
  Students' mindfulness will be evaluated with the Child and Adolescent Mindfulness Measure (La Greco et al., 2011), a 10-item self-report measure. Items are rated on a 5-point Likert scale (0 = Never true, 4 = Always true). Higher scores indicate greater mindfulness (range 0-40).
Self-Compassion | 10 days before intervention and 10 days after intervention
  Students' self-compassion will be assessed using the Self-Compassion Scale for Children (SCS-C; Sutton et al., 2018), a 12-item self-report measure. Items are rated on a 5-point Likert scale (1 = Almost never, 5 = Almost always). Higher scores indicate higher levels of self-compassion.
Self-Esteem | 10 days before intervention and 10 days after intervention
  Students' self-esteem will be assessed using the Rosenberg Self-Esteem Scale (Rosenberg, 1965), a 10-item self-report measure. Likert scale (0 = Strongly Disagree, 3 = Strongly Agree). Higher scores indicate higher self-esteem (range 0-30).
Executive functions - Visual Attention (NEPSY-II) | 10 days before intervention and 10 days after intervention
  Visual attention is assessed using the Visual Attention subtest of NEPSY-II, measuring speed and accuracy of visual attention. Low scores suggest deficits in selective attention or processing speed. The completion time is 180 seconds and accuracy is measured as the difference between the target stimuli identified and the distractor stimuli. The score is converted into scalar scores (minimum: 1 - maximum 19).
Executive functions - Working Memory (WISC-IV) | 10 days before intervention and 10 days after intervention
  Working memory/sequencing ability is assessed using the Letter-Number Sequencing subtest of WISC-IV. Scoring involves giving points for correctly sequenced items, leading to a raw score, which is then converted into a standardized scaled score (from 1 to 19) for comparison, reflecting the child's ability in short-term auditory memory and mental flexibility.
Executive functions - Inhibition Accuracy (TeleFE) | 10 days before intervention and 10 days after intervention
  Response inhibition is assessed using the Go/No-Go task from the TeleFE battery. The child is presented with a target stimulus and a non-target stimulus sequentially on the screen and must press the spacebar as soon as possible when the target stimulus appears. The task consists of 4 blocks, each with 35 target stimuli and 15 non-target stimuli. Each block therefore, contains a total of 50 stimuli (35 Go and 15 No-Go). In the present study, only the geometric shapes version of the Go/No-Go task was administered. From this task, an index of inhibition accuracy, calculated as the number of correct responses to non-target stimuli and expressed in percentiles (minimum: 0; maximum: 100), is obtained.
Executive functions - Inhibition Speed (TeleFE) | 10 days before intervention and 10 days after intervention
  Response inhibition is assessed using the Go/No-Go task from the TeleFE battery. The child is presented with a target stimulus and a non-target stimulus sequentially on the screen and must press the spacebar as soon as possible when the target stimulus appears. The task consists of 4 blocks, each with 35 target stimuli and 15 non-target stimuli. Each block therefore, contains a total of 50 stimuli (35 Go and 15 No-Go). In the present study, only the geometric shapes version of the Go/No-Go task was administered. From this task, an index of inhibition speed, calculated as the time of correct responses to target stimuli and expressed in percentiles (minimum: 0; maximum: 100), is obtained.
Executive functions - Interference control Accuracy (TeleFE) | 10 days before intervention and 10 days after intervention
  Interference control is assessed using the the 1st and 2nd blocks of the Flanker task from the TeleFE battery. The child is presented with a series of five arrows aligned on the screen, which can point all to the right or to the left (congruent condition), as well as the arrow in the middle can have the opposite direction to those on the side (incongruent condition). This task requires the child to rapidly shift between response criteria and implement them accurately. In all trials, a fixation point is displayed on the screen for approximately 600-1200 ms before each set of arrows. From this task, an accuracy index expressed in percentiles (minimum: 0; maximum: 100) from the correct responses of the first two blocks is obtained.
Executive functions - Interference control Speed (TeleFE) | 10 days before intervention and 10 days after intervention
  Interference control is assessed using the the 1st and 2nd blocks of the Flanker task from the TeleFE battery. The child is presented with a series of five arrows aligned on the screen, which can point all to the right or to the left (congruent condition), as well as the arrow in the middle can have the opposite direction to those on the side (incongruent condition). This task requires the child to rapidly shift between response criteria and implement them accurately. In all trials, a fixation point is displayed on the screen for approximately 600-1200 ms before each set of arrows. From this task, a speed index expressed in percentiles (minimum: 0; maximum: 100) from the reaction time at the correct response of the first two blocks is obtained.
Executive functions in daily life (QUFE) | 10 days before intervention and 10 days after intervention
  Executive function in daily life is assessed using the QUFE parent-report questionnaire, covering multiple aspects of executive functioning. Questionnaires for Executive Functions (QUFE; Schweiger & Marzocchi, 2008) for parents are completed to assess child's executive functioning within life context, specifically the home. The questionnaire consisted of 32 items on a five-point Likert scale, concerning 5 areas of investigation (cognitive self-regulation, behavioral self-regulation, material management, flexibility of adaptation, and spirit of initiative) for parents. A Global score is calculated (maximum: 160; minimum score: 32).
Emotional Instability | 10 days before intervention and 10 days after intervention
  Students' emotional instability is assessed using the parent-report Emotional Instability Scale (Pastorelli et al., 1997). This 20-item scale measures difficulties in emotion regulation and the tendency to experience negative affect. Answers are rated on a 3-point Likert scale (3 = Often, 2 = Sometimes, 1 = Never). Higher scores indicate higher emotional instability
Prosocial Behavior | 10 days before intervention and 10 days after intervention
  Students' prosocial behavior is assessed using the parent-report Prosocial Behavior Scale (Pastorelli et al., 1997). This 15-item scale evaluates positive social behaviors. Answers are rated on a 3-point Likert scale (3 = Often, 2 = Sometimes, 1 = Never). Higher scores indicated higher levels of prosociality.
Executive functions - Cognitive Flexibility Accuracy (TeleFE) | 10 days before intervention and 10 days after intervention
  Cognitive flexibility is assessed using the the 3rd block of the Flanker task from the TeleFE battery. The child is presented with a series of five arrows aligned on the screen, which can point all to the right or to the left (congruent condition), as well as the arrow in the middle can have the opposite direction to those on the side (incongruent condition). This task requires the child to rapidly shift between response criteria and implement them accurately. In all trials, a fixation point is displayed on the screen for approximately 600-1200 ms before each set of arrows. From this task, an accuracy index expressed in percentiles (minimum: 0; maximum: 100) from the correct responses of the third is obtained.
Executive functions - Cognitive Flexibility Speed (TeleFE) | 10 days before intervention and 10 days after intervention
  Cognitive flexibility is assessed using the the 3rd block of the Flanker task from the TeleFE battery. The child is presented with a series of five arrows aligned on the screen, which can point all to the right or to the left (congruent condition), as well as the arrow in the middle can have the opposite direction to those on the side (incongruent condition). This task requires the child to rapidly shift between response criteria and implement them accurately. In all trials, a fixation point is displayed on the screen for approximately 600-1200 ms before each set of arrows. From this task, a speed expressed in percentiles (minimum: 0; maximum: 100) from the reaction time of correct responses of the third block is obtained.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Università degli Studi di Firenze, Dipartimento di Scienze della Formazione e Psicologia, Florence, Firenze
  - Università di Pisa, Pisa, Pisa
  - IRCCS Fondazione Stella Maris, Pisa, Pisa
  - John Cabot University, Roma, Roma